CLINICAL TRIAL: NCT05984498
Title: An Investigation of the Physiological and Psychosocial Mechanisms Underpinning Balance Impairment in People With Chronic Obstructive Pulmonary Disease
Brief Title: Understanding Balance Impairment in COPD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Teesside University (Other)
Responsible Party: Principal Investigator, Samantha Harrison, Professor of Respiratory Rehabilitation, Teesside University
Other Study IDs: 2022 Aug 10959 Harrison; NIHR300856 (Other Grant/Funding Number: National Institute of Health Research (UK))
Record Dates: First submitted 2023-07-21; First posted 2023-08-09 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-08

CONDITIONS: Chronic Obstructive Pulmonary Disease; Healthy Volunteers
Keywords: Chronic, Obstructive Pulmonary Disease; Balance; Falls; Nerve Function; Muscle Function; Lived Experience
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COPD group: People with a spirometry confirmed diagnosis of Chronic Obstructive Pulmonary Disease (COPD)
- Healthy Controls: Older adults over the age of 55 who do not have COPD

SUMMARY:
This study is an observational study investigating the mechanisms of balance problems in people with COPD and how COPD impacts them living their daily lives.

The main objectives of this study are:

* To quantify the relationship between balance and aspects of neuromuscular function in individuals with COPD, and compared to age-matched healthy controls
* To understand the lived experience of people with COPD and their carers

Participants will attend an appointment at the University rehab lab to:

* Complete a balance test
* Fill out some questionnaires on mood, health status and balance and falls
* Complete some walking tests
* Have their body composition measured
* Have the function and strength of their leg nerves and muscles tested Researchers will compare people with COPD and healthy controls (older adults without COPD or other conditions known to impact balance) to see if any of the things measured are impacting the balance of people with COPD more than their peers without COPD.
* For 10 people with COPD only they will be visited at home to observe how they carry out everyday tasks and 5 of those 10 will have a follow up interview.

Researchers will take notes and record interviews and look for similarities and interesting points in the notes and transcripts of the interviews to build a picture of what living with COPD is like.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is a progressive condition that affects around 1.2million people in the UK. Breathlessness is the main symptom but people with COPD are also more likely to fall than healthy people of the same age. Falling has emotional consequences, such as feelings of shame, embarrassment and fear of falling in public which leads to avoidance of outdoor activities. Researchers do not know why people with COPD fall more but they have poor balance which may, in part, be due to problems with sensory and muscle responses that would usually maintain balance. Symptoms of breathlessness and pain, plus inactivity, may further impact balance. Physical and social environments may also have a role in falls risk, but this has yet to be investigated. Pulmonary Rehabilitation (PR) which includes stamina and strength exercises, alongside education and emotional support is standard treatment for COPD but it does not include any balance exercises, meaning people with COPD who are at a greater risk of falling do not receive any routine treatment to improve balance. This study aims to investigate the physical, psychological, social and environmental factors impacting on balance in people with COPD by comparing them to older adults without COPD. The study will recruit from local hospital services (people with COPD and their carers without COPD) and within the community (healthy older adults). Balance, muscle function (size, strength and speed of nerve conduction) and physical activity will be measured, and the two groups compared. Researchers will also observe patients in their own homes and do follow up interviews to understand what it is like to live with COPD and the challenges people face. The information from this study will be used in conjunction with stakeholders to co design an intervention to improve balance in people with COPD.

ELIGIBILITY:
Inclusion Criteria:

COPD

* Have a spirometry confirmed diagnosis of COPD as per GOLD guidelines
* Stable COPD (six weeks clear of exacerbation)
* 55 years or over at the point of recruitment
* Able to communicate with good verbal English or use adaptive equipment to communicate
* Male or female Controls
* Free from a diagnosis of COPD (confirmed by spirometry)
* 55 years or over at the point of recruitment
* Able to communicate with good verbal English or use adaptive equipment to
* Communicate
* Male or female

Exclusion Criteria:

COPD

* Recent exacerbation of COPD (within the last six weeks)
* Under 55 years of age at the point of recruitment
* Any neurological or musculoskeletal diagnoses (e.g., strokes, Parkinson's disease or chronic pain that interferes with ability to safely complete the tests
* Unable to provide written informed consent
* Unable to speak English or no translation options available
* Diagnosed but not corrected visual, vestibular disturbance and peripheral neuropathy
* Vasovagal syncope
* Not independent living (e.g., living in a care home or prison) Controls
* Abnormal lung function (FEV1 and FVC equal to or greater than 80% and FEV1/FVC equal to greater than 70%)
* Under 55 years of age at the point of recruitment
* Any neurological or musculoskeletal impairment that would significantly affect balance impacting ability to safely complete the assessments
* Unable to provide written informed consent
* Unable to speak English or no translation options available
* Any uncorrected visual or somatosensory disturbance
* Vasovagal syncope
* Living in a care home or in prison

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: People living with COPD and people without COPD living in community settings in the North East of England, UK
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-07-17 (Actual); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Balance Evaluation Systems Test (BESTest) | baseline only
  27 functional tasks scored on a 0-3 scale to give an overall percentage out from a maximum of 108 points. Higher scores indicate better balance.

SECONDARY OUTCOMES:
The Activities- Specific Balance Confidence Scale (ABC) | baseline only
  A questionnaire that assesses confidence for performing 16 activities without a loss of balance. Scores for each item range between 0 (not confident) and 100% (completely confident). The total score for each item is divided by the number of items (16).
The Elderly Falls Screening Test | baseline only
  A questionnaire and test that involves three questions relating to falls history in the previous 12-months and a gait speed and pattern assessment over a 5-meter course to establish falls risk. Score out of 5 with higher scores indicating a greater risk of falls.
Incremental Shuttle Walk Test | baseline only
  A walking test where participants walk between two cones that are 10 meters apart to a increasingly frequent paced beep to measure exercise capacity. The diatnace walked is reported to the nearest 10m.
COPD Assessment Test | baseline only
  A questionnaire measuring COPD health related quality of life. Scored between 0 and 40 with higher scores indicating the greatest impact of COPD on quality of life.
Medical Research Council Dyspnoea Scale | baseline only
  A one question scale (0-4) of the impact of breathlessness with higher scores indicating greater impact of symptoms.
Lung function testing (spirometry) Forced expiratory volume in one second (FEV1) and FEV1/forced vital capacity (FEV1/FVC) | baseline only
  A measure of lung function used to define COPD. Participants blow into a handheld spirometry device. FEV1 and FEV1 / FVC will be recorded.
Patient Health Questionnaire-9 (depression) | baseline only
  A one page questionnaire that measures symptoms of depression and low mood. Scored out of 27 with higher scores indicated greater symptoms of depression.
Generalised Anxiety Disorder-7 Questionnaire (anxiety) | baseline only
  A one page questionnaire that measures symptoms of anxiety. Scored out of 21 with higher scores indicating worse symptoms of depression.
Brief Pain Inventory | baseline only
  A two page questionnaire that records pain, pain intensity, pain location and pain interference. It consists of 9 items which are rated 0-10 with higher scores indicating a greater severity of pain.
Somatosensory accuracy | baseline only
  Vibration sensation perception will be measured with a neurothesiometer device on both big toes.
Maximal Voluntary Contraction Strength | baseline only
  The maximal strength that participants can generate in their thigh and calf muscles will be measured with a biodex dynamometer
Voluntary Activation Test | baseline only
  The amount of muscle available on top of a voluntary contraction in the quadriceps muscle will be measured using the biodex dynamometer and an electrical stimulus over the thigh muscles (Interpolated Twitch Technique)
Hoffman's Reflex | baseline only
  The speed and size of nerve response to a stimulus that mimics balance reactions will be measured in the tibial nerve by placing a small bar over the back of the knee that gives an electrical stimulus to the nerve.
Maximum grip strength | baseline only
  Participants hold a handheld dynamometer in their hands and squeeze the device to measure grip strength.
Physical Activity Monitor | baseline through to 7 days
  Participants will be asked to wear a watch sized device (Actigraph Physical Activity Monitor) on their wrists for 7 days. The actigraph device measures levels of physical activity
EuroQOL-5D-5Level | baseline only
  The EQ-5D-5L descriptive system comprises five dimensions (MOBILITY, SELF-CARE, USUAL ACTIVITIES, PAIN /DISCOMFORT and ANXIETY / DEPRESSION) and each dimension has five response levels (no problems to unable/severe problems). Responses form a 5 digit code.
  no problems, slight problems, moderate problems, severe problems, unable to /extreme problems.
Bioelectrical impendence analysis to record whole body composition of muscle, bone and fat | baseline only
  A bioelectrical impedance device (Tanita BIA) will record measures of body composition

CONTACTS AND LOCATIONS:
Overall Officials: Samantha L Harrison, PhD, Study Chair — Teesside University
Locations (1):
- Teesside University, Middlesbrough, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided